CLINICAL TRIAL: NCT01783886
Title: A Randomized, Double Masked, Active Controlled, Phase III Study of the Efficacy and Safety of Repeated Doses of Intravitreal VEGF Trap Eye in Subjects With Diabetic Macular Edema
Brief Title: Efficacy and Safety of VEGF Trap Eye in Diabetic Macular Edema (DME) With Central Involvement
Acronym: VIVID EAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15161
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Macular Edema
Keywords: Diabetic Macular Edema; DME; VEGF Trap-Eye; best-corrected visual acuity (BCVA)
MeSH Terms: conditions — Macular Edema | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravitreal Aflibercept Injection 2Q4 (Experimental): Participants received 2 mg Intravitreal aflibercept injection (IAI) (Eylea, VEGF [vascular endothelial growth factor] Trap-Eye, BAY86-5321) every 4 weeks (2Q4) over 48 weeks.
  Interventions: Biological: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Intravitreal Aflibercept Injection 2Q8 (Experimental): Participants received 2 mg Intravitreal aflibercept injection (IAI) (Eylea, VEGF Trap-Eye, BAY86-5321) every 4 weeks until Week 16 and every 8 weeks (2Q8) thereafter, over 48 weeks.
  Interventions: Biological: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Macular Laser Photocoagulation (Active Comparator): Participants received laser treatment at baseline and as needed at visits at which laser retreatment criteria were met, but no more frequently than every 12 weeks over 48 weeks.
  Interventions: Procedure: Macular Laser Photocoagulation

INTERVENTIONS:
Biological: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Participants received 2mg Intravitreal aflibercept injection (IAI) (EYLEA, VEGF Trap-Eye, BAY86-5321) every 4 weeks (2Q4).
  Arms: Intravitreal Aflibercept Injection 2Q4
Biological: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Participants received 2mg Intravitreal aflibercept injection (IAI) (EYLEA, VEGF Trap-Eye, BAY86-5321) every 4 weeks for 5 visits followed by injections every 8 weeks (2Q8).
  Arms: Intravitreal Aflibercept Injection 2Q8
Procedure: Macular Laser Photocoagulation — Participants received laser treatment at baseline and as needed at visits at which laser retreatment criteria were met, but no more frequently than every 12 weeks.
  Arms: Macular Laser Photocoagulation

SUMMARY:
To determine the efficacy of intravitreally (IVT) administered VEGF Trap-Eye on the best-corrected visual acuity (BCVA) assessed by the early treatment diabetic retinopathy study (ETDRS) chart in subjects with diabetic macular edema (DME) with central involvement.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years with type 1 or 2 diabetes mellitus
* Subjects with diabetic macular edema (DME) secondary to diabetes mellitus involving the center of the macula in the study eye
* Decrease in vision determined to be primarily the result of DME in the study eye
* Best-corrected visual acuity (BCVA) early treatment diabetic retinopathy study (ETDRS) letter score of 73 to 24 (20/40 to 20/320) in the study eye

Exclusion Criteria:

* Laser photocoagulation (panretinal or macular) in the study eye within 90 days of Day 1
* More than 2 previous macular laser treatments in the study eye
* Previous use of intraocular or periocular corticosteroids in the study eye within 120 days of Day 1
* Previous treatment with antiangiogenic drugs in either eye (pegaptanib sodium, bevacizumab, ranibizumab etc.) within 90 days of Day 1
* Active proliferative diabetic retinopathy (PDR) in the study eye
* Uncontrolled diabetes mellitus, as defined by HbA1c >12%
* Only 1 functional eye even if that eye is otherwise eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- China (13):
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Changsha, Hunan
  - Shenyang, Liaoning
  - Xi'an, Shaanxi
  - Qingdao, Shandong
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- Hong Kong (2):
  - Hong Kong
  - Kowloon
- Russia (3):
  - Moscow
  - Novosibirsk
  - Saint Petersburg
- Seoul, South Korea

REFERENCES:
- [Derived] Chen YX, Li XX, Yoon YH, Sun X, Astakhov Y, Xu G, Wang H, Ren X, Asmus F; VIVID-East investigators. Intravitreal Aflibercept versus Laser Photocoagulation in Asian Patients with Diabetic Macular Edema: The VIVID-East Study. Clin Ophthalmol. 2020 Mar 9;14:741-750. doi: 10.2147/OPTH.S235267. eCollection 2020. PMID 32210527
- [Derived] Ming J, Zhang Y, Xu X, Zhao M, Wang Y, Chen Y, Zhang F, Wang J, Liu J, Zhao X, Han R, Hu S. Cost-effectiveness analysis of intravitreal aflibercept in the treatment of diabetic macular edema in China. J Comp Eff Res. 2020 Feb;9(3):161-175. doi: 10.2217/cer-2019-0174. Epub 2020 Jan 6. PMID 31904267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at centers in China, Hong Kong, South Korea, and Russian Federation between 18 February 2013 (first participant first visit) and 09 March 2015 (last participant last visit) (data cut-off date).
Pre-assignment Details: Overall 539 participants were screened, of them 381 participants were randomized, and 378 participants were allocated to treatment.
Groups:
- Intravitreal Aflibercept Injection 2Q4: Participants received 2 milligram (mg) Intravitreal aflibercept injection (IAI) (Eylea, VEGF [vascular endothelial growth factor] Trap-Eye, BAY86-5321) every 4 weeks (2Q4) over 48 weeks.
Period: Overall Study
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Started | 127 | 127 | 127
Participants Received Treatment | 127 | 127 | 124
Completed | 122 | 116 | 117
Not Completed | 5 | 11 | 10
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Protocol deviation | 0 | 0 | 2
Not completed — Withdrawal of consent by participant | 1 | 3 | 4
Not completed — Adverse Event | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Intravitreal Aflibercept Injection 2Q4: Participants received 2 mg Intravitreal aflibercept injection (IAI) (Eylea, VEGF [vascular endothelial growth factor] Trap-Eye, BAY86-5321) 2Q4 over 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation | Total
Number analyzed (Participants) | 127 | 127 | 124 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.3) | 57.6 (10.1) | 58.8 (10.5) | 58.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 60 | 60 | 188
  Male | 59 | 67 | 64 | 190
Region of Enrollment [Number; unit: participants] — Geographic region
  participants
    China | 101 | 101 | 99 | 301
    Russia | 10 | 10 | 9 | 29
    Other Asia-Pacific (Hong Kong, Korea) | 16 | 16 | 16 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 52 - Last Observation Carried Forward (LOCF)
Description: Visual function of the study eye was assessed using the ETDRS protocol, which is a widely accepted international standard for macular laser photocoagulation treatment. A higher score represents better functioning. LOCF censored measurements after additional treatment.
Time Frame: Baseline up to week 52
Population: Full analysis set (FAS) included all randomized participants who received any study treatment, had a baseline measurement of BCVA, and had at least 1 post-baseline assessment of BCVA. FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Number analyzed (Participants) | 127 | 126 | 124
Letters correctly read | 13.7 (8.4) | 12.8 (9.5) | -0.2 (13.5)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 14.1, 97.5% CI 2-sided [10.9 to 17.2] — Least Square (LS) mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 13.6, 97.5% CI 2-sided [10.2 to 16.9] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser

2. Secondary Outcome: Percentage of Participants Who Gained at Least 10 Letters in BCVA as Measured by ETDRS Letter Score Compared With Baseline at Week 52 - LOCF
Description: Visual function of the study eye was assessed using the ETDRS protocol. A higher score represents better functioning.
Time Frame: Baseline up to week 52
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Number analyzed (Participants) | 127 | 126 | 124
Percentage of participants | 70.9 | 62.7 | 23.4
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted difference = 47.4, 97.5% CI 2-sided [35.0 to 59.9] — Cochran-Mantel-Haenszel (CMH). The estimate is calculated as EYLEA minus Laser
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted difference = 39.2, 97.5% CI 2-sided [26.3 to 52.1] — The estimate is calculated as EYLEA minus Laser

3. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters in BCVA as Measured by ETDRS Letter Score Compared With Baseline at Week 52 - LOCF
Description: Visual function of the study eye was assessed using the ETDRS protocol. A higher score represents better functioning.
Time Frame: Baseline up to week 52
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Number analyzed (Participants) | 127 | 126 | 124
Percentage of participants | 43.3 | 36.5 | 12.1
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted difference = 31.1, 97.5% CI 2-sided [19.2 to 43.0] — The estimate is calculated as EYLEA minus Laser
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted difference = 24.3, 97.5% CI 2-sided [12.6 to 35.9] — The estimate is calculated as EYLEA minus Laser

4. Secondary Outcome: Percentage of Participants With a Greater Than Equal (>=) Two-step Improvement From Baseline in the ETDRS Diabetic Retinopathy Severity Score (DRSS) as Assessed by Fundus Photography (FP) at Week 52 - LOCF
Description: ETDRS DRSS: None (level 10); Mild to moderate nonproliferative diabetic retinopathy (DR) (levels 14, 15, 20, 35, and 43); Moderately severe/severe nonproliferative DR (levels 47 and 53); Mild/moderate/high-risk/advanced proliferative DR (levels 61, 65, 71,75, 81, and 85)
Time Frame: Baseline up to week 52
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Number analyzed (Participants) | 122 | 122 | 120
Percentage of participants | 60.7 | 62.3 | 21.7
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted difference = 39.1, 97.5% CI 2-sided [26.0 to 52.2] — The estimate is calculated as EYLEA minus Laser
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted difference = 40.6, 97.5% CI 2-sided [27.6 to 53.7] — The estimate is calculated as EYLEA minus Laser

5. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) at Week 52 as Assessed on Optical Coherence Tomography (OCT) - LOCF
Description: CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from Baseline indicated improvement.
Time Frame: Baseline up to week 52
Population: FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Number analyzed (Participants) | 126 | 126 | 124
micrometer | -238.7 (172.5) | -234.7 (160.8) | -109.3 (206.9)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, ANCOVA; Median Difference (Final Values) = -130.5, 97.5% CI 2-sided [-171.2 to -89.9] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -131.4, 97.5% CI 2-sided [-172.8 to -89.9] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser

6. Secondary Outcome: Change From Baseline in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Near Activities Subscale at Week 52 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales that are all scored from 0-100. Near activities are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf.
Time Frame: Baseline up to week 52
Population: FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Number analyzed (Participants) | 124 | 122 | 119
Scores on a scale | 6.65 (23.86) | 7.28 (22.95) | 0.04 (24.39)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p = 0.0364, ANCOVA; Mean Difference (Final Values) = 5.78, 97.5% CI 2-sided [-0.41 to 11.97] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p = 0.0113, ANCOVA; Mean Difference (Final Values) = 6.87, 97.5% CI 2-sided [0.80 to 12.94] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser

7. Secondary Outcome: Change From Baseline in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Distance Activities Subscale at Week 52 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales that are all scored from 0-100. Distance activities are defined as reading street signs or names on stores, and going down stairs, steps, or curbs.
Time Frame: Baseline up to week 52
Population: FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Number analyzed (Participants) | 124 | 122 | 119
Scores on a scale | 3.93 (22.36) | 10.25 (21.44) | 0.04 (23.14)
Statistical Analysis 1: Comparison: Intravitreal Aflibercept Injection 2Q4 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p = 0.2688, ANCOVA; Mean Difference (Final Values) = 2.81, 97.5% CI 2-sided [-2.90 to 8.53] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser
Statistical Analysis 2: Comparison: Intravitreal Aflibercept Injection 2Q8 vs Macular Laser Photocoagulation; Test type: Superiority or Other; p = 0.0009, ANCOVA; Mean Difference (Final Values) = 8.01, 97.5% CI 2-sided [2.64 to 13.37] — LS mean difference from ANCOVA. The estimate is calculated as EYLEA minus Laser

ADVERSE EVENTS:
Time Frame: From the start of study treatment up to 52 weeks
Arm/Group | Intravitreal Aflibercept Injection 2Q4 | Intravitreal Aflibercept Injection 2Q8 | Macular Laser Photocoagulation
Serious Adverse Events (participants affected / at risk) | 19/127 | 22/127 | 24/124
Other Adverse Events (participants affected / at risk) | 87/127 | 83/127 | 89/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Aflibercept Injection 2Q4 (N=127) | Intravitreal Aflibercept Injection 2Q8 (N=127) | Macular Laser Photocoagulation (N=124)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 2 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 2
Hyphaema (Eye disorders) | 0 | 0 | 1
Papilloedema (Eye disorders) | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 2
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 4
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Dacryocystitis (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Renal osteodystrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant lymphoid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 2 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 2
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Aflibercept Injection 2Q4 (N=127) | Intravitreal Aflibercept Injection 2Q8 (N=127) | Macular Laser Photocoagulation (N=124)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 7
Conjunctival haemorrhage (Eye disorders) | 18 | 13 | 6
Diabetic retinal oedema (Eye disorders) | 17 | 13 | 15
Diabetic retinopathy (Eye disorders) | 5 | 7 | 7
Macular fibrosis (Eye disorders) | 6 | 7 | 4
Macular oedema (Eye disorders) | 8 | 10 | 9
Retinal aneurysm (Eye disorders) | 9 | 13 | 10
Retinal exudates (Eye disorders) | 8 | 13 | 5
Retinal haemorrhage (Eye disorders) | 14 | 17 | 12
Vision blurred (Eye disorders) | 4 | 7 | 3
Visual acuity reduced (Eye disorders) | 12 | 14 | 24
Vitreous haemorrhage (Eye disorders) | 4 | 3 | 7
Conjunctivitis (Infections and infestations) | 8 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 8 | 9 | 7
Glycosylated haemoglobin increased (Investigations) | 5 | 9 | 5
Visual acuity tests abnormal (Investigations) | 9 | 3 | 15
Diabetes mellitus (Metabolism and nutrition disorders) | 12 | 10 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 3
Hypertension (Vascular disorders) | 10 | 15 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.